CLINICAL TRIAL: NCT03469453
Title: Internet-delivered Cognitive Behavioral Therapy for Adolescents With Generalized Anxiety Disorder - a Multiple Baseline Evaluation
Brief Title: Internet-delivered CBT for Adolescents With GAD
Acronym: BIPWorry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Serlachius, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN DNR 2017/1879-31/5
Record Dates: First submitted 2017-12-20; First posted 2018-03-19 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; Adolescents; Internet-delivered Cognitive behavioral therapy; ICBT; CBT
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered CBT (Experimental): Internet-delivered Cognitive Behavioral Therapy (ICBT) for GAD, 10 weeks. Patients and their parents work with separate programs via the Internet. Both have contact with a therapist. Participants practice awareness of worry through daily worry monitoring. They identify their own behaviors that reinforce worry, i.e. control and avoidance behaviors. The program gives a rationale for behavior change, which is then implemented. Participants practice problem solving and exposure to uncertainty inducing situations and thoughts. Parents receive support and psycho education about worry. They practice alternative parental behaviors, which decrease focus on worry while validating the child's feelings. Treatment contains planning for maintenance of treatment gains for both patients and parents.
  Interventions: Behavioral: Internet-Delivered Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Internet-Delivered Cognitive Behavioral Therapy — Therapist-supported CBT delivered online.
  Other Names: ICBT

SUMMARY:
This multiple baseline evaluation aims to test the feasibility and preliminary effectiveness of Internet-delivered cognitive behavioral therapy (ICBT) for adolescents with Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
This pilot study aims to test Internet-delivered Cognitive Behavioral Therapy (ICBT) for adolescents with Generalized Anxiety Disorder (GAD)

The study has a single case research design (multiple baseline) and will include 12 participants with GAD according to a semi structured diagnostic interview.

Participants will be randomized to either two, six or ten weeks baseline measurements prior to starting treatment, and will thus work as their own controls.

Primary outcome measures will be collected at 10 weeks after treatment start. Follow-up assessments will be made three month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* A score on the Penn State Worry Questionnaire for Children (PSWQ-C) of > 30
* Fulfilling DSM-5 criteria for Generalized Anxiety Disorder
* No other disorder or symptoms present in need of more urgent treatment
* Aged between 13 and 17 years
* Ability to read and write in Swedish
* A parent or caregiver that is able to participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment
* No other ongoing psychological treatment for any disorder

Exclusion Criteria:

* The presence of symptoms suggestive of a current diagnosis of Autistic Spectrum Disorder, Schizophrenia, Bipolar Disorder, Anorexia Nervosa, Bulimia, or Substance Use Disorder
* Present risk of suicide
* Present occurrence of domestic violence
* Completed CBT for any anxiety disorder within the last 6 months (defined as at least 5 sessions of CBT including in vivo exposure sessions)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Brief Penn State Worry Questionnaire for Children | 10 weeks after baseline
  Self-assessment of excessive worry for individual analysis in multiple baseline evaluation
Penn State Worry Questionnaire for Children | 10, 14 and 22 weeks after baseline
  Child and parent version, lower values indicating decrease in worry. Assessments used in group statistical analysis of clinical outcome

SECONDARY OUTCOMES:
Brief Intolerance of Uncertainty Scale | 10, 14 and 22 weeks after baseline
  Child version, lower values indicating decrease in intolerance of uncertainty
Brief Cognitive Avoidance Questionnaire | 10, 14 and 22 weeks after baseline
  Child version, lower values indicating decrease in cognitive avoidance
Negative Problem Orientation Questionnaire, abbreviated | 10, 14 and 22 weeks after baseline
  Child version, lower values indicating decrease in negative problem orientation
Revised Children's Anxiety and Depression Scale | 10, 14 and 22 weeks after baseline
  Child and parent versions, lower values indicating decrease in anxiety and depression
Education, Work and Social Adjustment Scale | 10 and 22 weeks after baseline
  Child and parent versions, , lower values indicating decreased impairment due to worry
Clinical Global Impression - Improvement | 10, 14 and 22 weeks after baseline
  Clinician rated, higher values indicate larger improvement after treatment
Anxiety Disorder Interview Schedule for the Diagnostic and Statistical Manual -IV | 10, 14 and 22 weeks after baseline
  Diagnostic interview
Clinician Severity Rating | 10, 14 and 22 weeks after baseline
  Clinician rated severity with lower values indicating lower level of severity of a disorder
Children's Global Assessment Scale | 10, 14 and 22 weeks after baseline
  Clinician rated global functioning, higher values indicate higher functioning

OTHER OUTCOMES:
Treatment credibility and expectancy scale (child and parent version) | 10 weeks after baseline
  A 5-item scale, rated from 0-10, with higher scores indicating higher treatment credibility and expectancy.
Negative Events Questionnaire (child and parent version) | 10 weeks after baseline
  The 5-item scale queries negative events during treatment and if the participants attributes the event to the intervention.
Client satisfaction questionnaire | 10 weeks after baseline
  Child- and parent rated treatment satisfaction is rated on an eight items scale,ange 0-3, with higher score indicating higher satisfaction..
Internet intervention Patient Adherence Scale | 5 and 10 weeks after baseline
  Clinician rated, 5-item scale ranging from 0-4 with higher scores indicating higher participant adherence to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No